CLINICAL TRIAL: NCT00002414
Title: Randomized, Double-Blind, Parallel Group, Placebo Controlled, Tolerability, Safety and Pilot Efficacy Study of CPI-1189 in HIV Infected Individuals With Cognitive and Motor Impairment
Brief Title: Safety and Effectiveness of Giving CPI-1189 to HIV-Infected Patients With AIDS Dementia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Centaur Pharmaceuticals (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 289B; CPI001189-ADC01
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2000-04

CONDITIONS: HIV Infections
Keywords: AIDS Dementia Complex; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections; AIDS Dementia Complex | interventions — CPI 1189

INTERVENTIONS:
Drug: CPI-1189

SUMMARY:
The purpose of this study is to see if it is safe and effective to give CPI-1189 to patients with AIDS dementia.

Advanced HIV infection can cause AIDS dementia (brain damage due to HIV leading to loss of memory and muscle control). CPI-1189 may be able to postpone AIDS dementia or slow it down.

DETAILED DESCRIPTION:
Late-stage HIV infection can cause AIDS dementia (brain damage due to HIV leading to loss of memory and muscle control). CPI-1189 may be able to postpone AIDS dementia or slow it down.

Patients are randomized to receive either placebo or one of two oral doses of CPI-1189 daily. Patients are assessed for safety and tolerability during Weeks 2, 6, and 10. At Week 10, efficacy assessments are also made. For those who volunteer, a sample of cerebrospinal fluid is obtained at baseline and at Week 10. Blood samples for CPI-1189 pharmacokinetic trough measurements are taken at Weeks 2 and 10. The open-label phase starts at Week 11. At Weeks 13 and 16, a safety evaluation is performed. At the end of the open-label phase, Week 22, a final set of safety and efficacy assessments and a blood sample for CPI-1189 pharmacokinetic trough measurement are obtained.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Are at least 18 years old.
* Have symptoms of AIDS dementia including forgetfulness, loss of concentration, slow mental processing, or a loss of muscle control.
* Have been on stable anti-HIV drug therapy for the past 6 weeks (if you are taking anti-HIV drugs).

Exclusion Criteria

You will not be eligible for this study if you:

* Have certain serious medical conditions, such as a mental disorder or an opportunistic (AIDS-related) infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60

CONTACTS AND LOCATIONS:
Overall Officials: Clifford DB, Study Chair
Locations (6):
- United States (6):
  - Alzheimers Disease Research Ctr 0948 / UCSD, San Diego, California
  - Northwestern Univ / Dept of Neurology, Chicago, Illinois
  - Johns Hopkins Hosp / Dept of Neurology / Meyer 6109, Baltimore, Maryland
  - Washington Univ Sch of Med / Dept of Neurology, St Louis, Missouri
  - Columbia Univ / Sergievsky Ctr Physicians and Surgeons, New York, New York
  - Univ of Rochester / Strong Memorial Hosp, Rochester, New York

REFERENCES:
- [Background] Clifford DB, McArthur JC, Schifitto G, Kieburtz K, McDermott MP, Letendre S, Cohen BA, Marder K, Ellis RJ, Marra CM; Neurologic AIDS Research Consortium. A randomized clinical trial of CPI-1189 for HIV-associated cognitive-motor impairment. Neurology. 2002 Nov 26;59(10):1568-73. doi: 10.1212/01.wnl.0000034177.47015.da. PMID 12451199